CLINICAL TRIAL: NCT00933777
Title: SORAVE-Sorafenib and Everolimus in Solid Tumors. A Phase I Clinical Trial to Evaluate the Safety of Combined Sorafenib and Everolimus Treatment in Patients With Relapsed Solid Tumors
Brief Title: SORAVE - Sorafenib and Everolimus in Solid Tumors
Acronym: SORAVE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Wolf, Prof. Dr., Lung Cancer Group Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SORAVE
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapy with everolimus and sorafenib (Experimental): Dose finding: Treatment with defined dose of sorafenib of 2x400 mg with increasing dose of everolimus (2.5 mg, 5 mg, 7.5 mg, 10 mg) Extension: Treatment with defined dose of sorafenib of 2x400 mg with everolimus 7.5 mg
  Interventions: Drug: Combination of sorafenib and everolimus

INTERVENTIONS:
Drug: Combination of sorafenib and everolimus — Dose finding: Treatment with defined dose of sorafenib of 2x400 mg with increasing dose of everolimus (2.5 mg, 5 mg, 7.5 mg, 10 mg) Extension: Treatment with defined dose of sorafenib of 2x400 mg with everolimus 7.5 mg
  Other Names: Nexavar, RAD001

SUMMARY:
Dose finding part: A phase I clinical trial to evaluate the safety of combined sorafenib and everolimus treatment in patients with relapsed solid tumors (finished).

Extension part:Treatment of non-small cell lung cancer (NSCLC) with KRAS mutation after ≥ 1st relapse (recruiting)

DETAILED DESCRIPTION:
Dose finding part: Patients will be recruited to receive combination of defined sorafenib dose (2x400mg) with increasing dose of everolimus (2.5mg, 5mg, 7.5mg, 10mg). There will be a run-in phase of 14 days of everolimus followed by combination sorafenib+everolimus starting from day 15. The combination will be continued as long as it is tolerated by the patient and the patient benefits from the treatment according to RECIST criteria. The maximal tolerated dose will be establish in 3+3 design. Patients will be recruited sequentially at least 14 days apart. The next dose level according to 3+3 design will be initiated if all patients on the previous dose level reach day 29.

Extension part: Patients will be treated with a dose of 7,5 mg Everolimus for 14 days (run-in phase) and sorafenib 2x 400 mg until progression

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors relapsed after and/or refractory to standard therapy (dose finding part), KRAS mutated NSCLC patients after ≥ 1st relapse for the extension phase
* ≥ 18 years of age
* Performance status ECOG 0-2
* Life expectancy of at least 12 weeks
* Subjects with at least one measurable (CT or MRI) lesion
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1,500 /mm3
  * Platelet count ≥ 100 000/µL
  * Total bilirubin ≤ 1,5x upper limit of normal (ULN)
  * ALT and AST ≤ 2,5x ULN (≤ 5x ULN for patients with liver involvement)
  * Alkaline phosphatase < 4x ULN
  * Potassium within normal limits (WNL) or correctable with supplements
  * Total calcium (corrected for serum albumin) WNL or correctable with supplements
  * Magnesium WNL or correctable with supplements
  * PT-INR/PTT < 1.5 x ULN [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists]
  * Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance (CrCl) ≥ 50 ml/min calculated by either Cockcroft-Gault or by 24 hours urine collection
* More than 14 days since previous systemic therapy, radiotherapy and surgery
* Negative urine or serum HCG in women of childbearing potential
* Signed and dated informed consent before the start of specific protocol procedures

Exclusion Criteria:

* Squamous cell carcinoma histology in non-small cell lung cancer
* History of cardiac disease: congestive heart failure > NYHA class 2; active Coronary Arterial Disease (CAD), (MI more than 6 months prior to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy (except, when controlled by beta blockers or digoxin) or uncontrolled hypertension; for Extension phase: Long QT-Syndrome
* Active skin, mucosa, ocular or GI disorders of grade > 1
* Uncontrolled diabetes
* ≥ grade 3 hypercholesterolemia/hypertriglyceridemia or ≥ grade 2 hypercholesterolemia / hypertriglyceridemia with history of CAD (despite lipid lowering treatment if given)
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus and sorafenib (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* History of HIV infection or previously sero-positive for the virus
* History of Hepatitis B or/and C or previously sero-positive for the Hepatitis B or/and C virus
* Leptomeningeal or uncontrolled brain metastases, including patients who continue to require glucocorticoids or intrathecal chemotherapy for brain or leptomeningeal metastases (documented by lumbar puncture)
* Treatment with any other investigational drugs within the previous 14 days
* Patients with seizure disorder requiring anti-epileptics
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Previous treatment with mTOR inhibitors and/or known hypersensitivity to mTOR inhibitors
* Past or current history of cancer other than the entry diagnosis EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry
* Any person being in an institution on assignment of the respective authority
* Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information
* Women who are pregnant or breast feeding, or women who are able to conceive and unwilling to practice an effective method of birth control (safe hormonal methods or/and barrier contraception) during study and 2 months after the last study drug intake

For Extension part:

* Patients with medication that prolongs QTc and cannot be withdrawn (if the QTc prolonging medication is withdrawn - there must be a time interval of at least 7 days before starting treatment with sorafenib, in case of amiodarone the time interval is at least 90 days)
* Testing for Hepatitis B is mandatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-07; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To define a feasible treatment schedule for the combination therapy with sorafenib and everolimus | July 2009 - December 2011

SECONDARY OUTCOMES:
To determine the maximum tolerated dose (MTDs) of everolimus in combination with 2 x 400 mg sorafenib daily | July 2009 - December 2011
To analyze pharmacokinetic (PK) profiles (AUC, Cmax) of sorafenib and everolimus during combination therapy | July 2009 - December 2012
To determine the safety profile of the combination therapy with sorafenib + everolimus | July 2009 - December 2012
To correlate KRAS-mutation status with treatment response (extension phase) | December 2011 - December 2012

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Wolf, MD, Prof., Principal Investigator — Lung Cancer Group Cologne, Center for Integrated Oncology, Dep.I of Internal Medicine, University Hospital Cologne, Germany
Locations (1):
- Center for Integrated Oncology, Dep.I of Internal Medicine, University Hospital Cologne, Cologne, Germany

REFERENCES:
- [Background] Escudier B, Eisen T, Stadler WM, Szczylik C, Oudard S, Siebels M, Negrier S, Chevreau C, Solska E, Desai AA, Rolland F, Demkow T, Hutson TE, Gore M, Freeman S, Schwartz B, Shan M, Simantov R, Bukowski RM; TARGET Study Group. Sorafenib in advanced clear-cell renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):125-34. doi: 10.1056/NEJMoa060655. PMID 17215530
- [Background] Herbst RS, Johnson DH, Mininberg E, Carbone DP, Henderson T, Kim ES, Blumenschein G Jr, Lee JJ, Liu DD, Truong MT, Hong WK, Tran H, Tsao A, Xie D, Ramies DA, Mass R, Seshagiri S, Eberhard DA, Kelley SK, Sandler A. Phase I/II trial evaluating the anti-vascular endothelial growth factor monoclonal antibody bevacizumab in combination with the HER-1/epidermal growth factor receptor tyrosine kinase inhibitor erlotinib for patients with recurrent non-small-cell lung cancer. J Clin Oncol. 2005 Apr 10;23(11):2544-55. doi: 10.1200/JCO.2005.02.477. Epub 2005 Mar 7. PMID 15753462
- [Background] O'Donnell A, Faivre S, Burris HA 3rd, Rea D, Papadimitrakopoulou V, Shand N, Lane HA, Hazell K, Zoellner U, Kovarik JM, Brock C, Jones S, Raymond E, Judson I. Phase I pharmacokinetic and pharmacodynamic study of the oral mammalian target of rapamycin inhibitor everolimus in patients with advanced solid tumors. J Clin Oncol. 2008 Apr 1;26(10):1588-95. doi: 10.1200/JCO.2007.14.0988. Epub 2008 Mar 10. PMID 18332470
- [Background] Atkins MB, Hidalgo M, Stadler WM, Logan TF, Dutcher JP, Hudes GR, Park Y, Liou SH, Marshall B, Boni JP, Dukart G, Sherman ML. Randomized phase II study of multiple dose levels of CCI-779, a novel mammalian target of rapamycin kinase inhibitor, in patients with advanced refractory renal cell carcinoma. J Clin Oncol. 2004 Mar 1;22(5):909-18. doi: 10.1200/JCO.2004.08.185. PMID 14990647
- [Background] Spira A, Ettinger DS. Multidisciplinary management of lung cancer. N Engl J Med. 2004 Jan 22;350(4):379-92. doi: 10.1056/NEJMra035536. No abstract available. PMID 14736930
- [Background] Tabernero J, Rojo F, Calvo E, Burris H, Judson I, Hazell K, Martinelli E, Ramon y Cajal S, Jones S, Vidal L, Shand N, Macarulla T, Ramos FJ, Dimitrijevic S, Zoellner U, Tang P, Stumm M, Lane HA, Lebwohl D, Baselga J. Dose- and schedule-dependent inhibition of the mammalian target of rapamycin pathway with everolimus: a phase I tumor pharmacodynamic study in patients with advanced solid tumors. J Clin Oncol. 2008 Apr 1;26(10):1603-10. doi: 10.1200/JCO.2007.14.5482. Epub 2008 Mar 10. PMID 18332469
- [Background] Stroobants S, Verschakelen J, Vansteenkiste J. Value of FDG-PET in the management of non-small cell lung cancer. Eur J Radiol. 2003 Jan;45(1):49-59. doi: 10.1016/s0720-048x(02)00282-6. PMID 12499064
- [Background] Strumberg D, Richly H, Hilger RA, Schleucher N, Korfee S, Tewes M, Faghih M, Brendel E, Voliotis D, Haase CG, Schwartz B, Awada A, Voigtmann R, Scheulen ME, Seeber S. Phase I clinical and pharmacokinetic study of the Novel Raf kinase and vascular endothelial growth factor receptor inhibitor BAY 43-9006 in patients with advanced refractory solid tumors. J Clin Oncol. 2005 Feb 10;23(5):965-72. doi: 10.1200/JCO.2005.06.124. Epub 2004 Dec 21. PMID 15613696
- [Background] Moore M, Hirte HW, Siu L, Oza A, Hotte SJ, Petrenciuc O, Cihon F, Lathia C, Schwartz B. Phase I study to determine the safety and pharmacokinetics of the novel Raf kinase and VEGFR inhibitor BAY 43-9006, administered for 28 days on/7 days off in patients with advanced, refractory solid tumors. Ann Oncol. 2005 Oct;16(10):1688-94. doi: 10.1093/annonc/mdi310. Epub 2005 Jul 8. PMID 16006586
- [Background] Cascone T, Gridelli C, Ciardiello F. Combined targeted therapies in non-small cell lung cancer: a winner strategy? Curr Opin Oncol. 2007 Mar;19(2):98-102. doi: 10.1097/CCO.0b013e328011beec. PMID 17272980
- See also: Related Info — http://www.cio-koeln-bonn.de